CLINICAL TRIAL: NCT04938453
Title: Relative Bioavailability of 100 mg Nintedanib (Ofev®) Given as Four Capsules of 25 mg Compared to One Capsule of 100 mg Following Oral Administration in Healthy Male Subjects (an Open-label, Randomised, Single-dose, Two-period, Two-sequence Crossover Study)
Brief Title: A Study in Healthy Men to Test Whether Four Capsules of 25 mg Nintedanib Are Taken up in the Body in the Same Way as One 100 mg Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1199-0463; 2021-001052-34 (EudraCT Number)
Record Dates: First submitted 2021-06-23; First posted 2021-06-24 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2022-08

CONDITIONS: Healthy
MeSH Terms: interventions — nintedanib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nintedanib 4 X 25 mg (T) then nintedanib 1 X 100 mg (R)) (Experimental): first test (T), then reference (R) treatment
  Interventions: Drug: nintedanib 25 mg; Drug: nintedanib 100 mg
- nintedanib 1 X 100 mg (R) then nintedanib 4 X 25 mg (T) (Experimental): first reference (R), then test (T) treatment
  Interventions: Drug: nintedanib 25 mg; Drug: nintedanib 100 mg

INTERVENTIONS:
Drug: nintedanib 25 mg — soft gelatin capsule
Drug: nintedanib 100 mg — soft gelatin capsule
  Other Names: Ofev®

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of 100 mg nintedanib given as four capsules of 25 mg nintedanib compared with one capsule of 100 mg nintedanib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase I trial to test the relative bioavailability of 100 milligram (mg) nintedanib (Ofev®) given as four capsules of 25 mg compared to one capsule of 100 mg following oral administration in healthy male subjects (an open-label, randomised, single-dose, two-period, two-sequence crossover study).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Nintedanib 1 X 100 mg (R) / Nintedanib 4 X 25 mg (T): On Day 1 of Period 1 participants were administered once 1 soft gelatin capsule of 100 milligram (mg) of nintedanib (reference treatment (R)) orally with 240 milliliter (mL) of water after breakfast.
  On Day 1 of Period 2 participants were administered one single intake of 4 soft gelatin capsules of 25 mg of nintedanib (total administered dose = 100 mg) (test treatment (T)) orally with 240 mL of water after breakfast.
  There was a washout period of at least 7 days between the treatments.
- Nintedanib 4 X 25 mg (T) / Nintedanib 1 X 100 mg (R): On Day 1 of Period 1 participants were administered one single intake of 4 soft gelatin capsules of 25 milligram (mg) of nintedanib (total administered dose = 100 mg) (test treatment (T)) orally with 240 milliliter (mL) of water after breakfast.
  On Day 1 of Period 2 participants were administered once 1 soft gelatin capsule of 100 mg of nintedanib (reference treatment (R)) orally with 240 mL of water after breakfast.
  There was a washout period of at least 7 days between the treatments.
Period: Period 1
Arm/Group | Nintedanib 1 X 100 mg (R) / Nintedanib 4 X 25 mg (T) | Nintedanib 4 X 25 mg (T) / Nintedanib 1 X 100 mg (R)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout Period 1
Arm/Group | Nintedanib 1 X 100 mg (R) / Nintedanib 4 X 25 mg (T) | Nintedanib 4 X 25 mg (T) / Nintedanib 1 X 100 mg (R)
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1
Period: Period 2
Arm/Group | Nintedanib 1 X 100 mg (R) / Nintedanib 4 X 25 mg (T) | Nintedanib 4 X 25 mg (T) / Nintedanib 1 X 100 mg (R)
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): TS included all subjects who were randomised and treated with at least 1 dose of the investigational medicinal product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib 1 X 100 mg (R) / Nintedanib 4 X 25 mg (T) | Nintedanib 4 X 25 mg (T) / Nintedanib 1 X 100 mg (R) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.2 (10.1) | 32.4 (7.8) | 33.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Nintedanib in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the nintedanib in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
Time Frame: For both arms: Within 3 hours (h) before and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h, 24 h, 34 h, 48 h and 72h after nintedanib administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): The PKS included all subjects in the TS who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he contributed only 1 PK parameter value for 1 period to the statistical assessment.
Measure: Geometric Least Squares Mean (Standard Error); unit: hours (h) *nanogram(ng)/milliliter (mL)
Groups:
- Nintedanib 1 X 100 mg (R): This arm includes all participants who were administered once 1 soft gelatin capsule of 100 milligram (mg) of nintedanib (reference treatment (R)) orally with 240 milliliter (mL) of water after breakfast.
- Nintedanib 4 X 25 mg (T): This arm includes all participants who were administered one single intake of 4 soft gelatin capsules of 25 mg of nintedanib (total administered dose = 100 mg) (test treatment (T)) orally with 240 milliliter (mL) of water after breakfast.
Arm/Group | Nintedanib 1 X 100 mg (R) | Nintedanib 4 X 25 mg (T)
Number analyzed (Participants) | 19 | 19
hours (h) *nanogram(ng)/milliliter (mL) | 150.65 (NA) — Standard error is actually adjusted geometric standard error. Adjusted geometric standard error=1.07. | 148.34 (NA) — Standard error is actually adjusted geometric standard error. Adjusted geometric standard error=1.07.
Statistical Analysis 1: Comparison: Nintedanib 1 X 100 mg (R) vs Nintedanib 4 X 25 mg (T); The statistical model used for the analysis of this primary endpoint was an analysis of variance (ANOVA) model on the logarithmic scale. This model included effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Other; Ratio of GLSMs (%) = 98.47, 90% CI 2-sided [90.87 to 106.69], Standard Error of Mean 13.9 — Ratio of Geometric Least Squares Means (GLSMs) was calculated as (GLSM of "nintedanib 4 X 25 mg")/(GLSM of "nintedanib 1 X 100 mg"). Standard error of the mean is actually intra-individual geometric coefficient of variation (gCV [%])

2. Primary Outcome: Maximum Measured Concentration of Nintedanib in Plasma (Cmax)
Description: Maximum measured concentration of nintedanib in plasma (Cmax) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Deviation); unit: nanogram (ng)/milliliter (mL)
Arm/Group | Nintedanib 1 X 100 mg (R) | Nintedanib 4 X 25 mg (T)
Number analyzed (Participants) | 19 | 19
nanogram (ng)/milliliter (mL) | 15.23 (NA) — Standard error is actually adjusted geometric standard error. Adjusted geometric standard error=1.11. | 15.27 (NA) — Standard error is actually adjusted geometric standard error. Adjusted geometric standard error=1.11.
Statistical Analysis 1: Comparison: Nintedanib 1 X 100 mg (R) vs Nintedanib 4 X 25 mg (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of GLSMs (%) = 100.29, 90% CI 2-sided [85.05 to 118.24], Standard Error of Mean 29.2 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Concentration-time Curve of Nintedanib in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of nintedanib in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hours * nanogram/milliliter
Arm/Group | Nintedanib 1 X 100 mg (R) | Nintedanib 4 X 25 mg (T)
Number analyzed (Participants) | 19 | 19
hours * nanogram/milliliter | 157.55 (NA) — Standard error is actually adjusted geometric standard error. Adjusted geometric standard error=1.07. | 155.85 (NA) — Standard error is actually adjusted geometric standard error. Adjusted geometric standard error=1.07.
Statistical Analysis 1: Comparison: Nintedanib 1 X 100 mg (R) vs Nintedanib 4 X 25 mg (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of GLSMs (%) = 98.92, 90% CI 2-sided [91.35 to 107.12], Standard Error of Mean 13.8 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: For both arms: From drug administration until 14 days thereafter.
Description: Treated set (TS): TS included all subjects who were randomised and treated with at least 1 dose of the investigational medicinal product.
Groups:
- Nintedanib 1 X 100 mg (R): This arm includes all participants who were administered once 1 soft gelatin capsule of of 100 milligram (mg) of nintedanib (reference treatment (R)) orally with 240 milliliter (mL) of water after breakfast.
Arm/Group | Nintedanib 1 X 100 mg (R) | Nintedanib 4 X 25 mg (T)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 10/19 | 5/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib 1 X 100 mg (R) (N=19) | Nintedanib 4 X 25 mg (T) (N=19)
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Macule (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT04938453/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT04938453/SAP_001.pdf